CLINICAL TRIAL: NCT06573502
Title: Assessment of Platelet Rich Plasma With Injectable Platelet Rich Fibrin VS Platelet Rich Plasma Vs Platelet Rich Fibrin in Management of Temporomandibular Joint Osteoarthritis
Brief Title: Platelet Rich Plasma Combined With Platelet Rich Fibrin in Management of Temporomandibular Joint Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aliaa Babekir Ahmed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Aliaa Babekir Ahmed Mohamed, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Not selected
Record Dates: First submitted 2024-07-31; First posted 2024-08-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide; Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- prp with prf group (Experimental): Pt will recievd prp with prf
  Interventions: Combination Product: Prp with prf or prp or prf
- prp group (Active Comparator): Pt will recieve prp only
  Interventions: Combination Product: Prp with prf or prp or prf
- prf group (Experimental): Pt will recieve prf only
  Interventions: Combination Product: Prp with prf or prp or prf

INTERVENTIONS:
Combination Product: Prp with prf or prp or prf — Combination

SUMMARY:
Studying effectiveness of prp with prf comparing with prp or prf for mangement of tmj osteoarthritis as result in pain and mandibular movement in adult pt

DETAILED DESCRIPTION:
45 pt assigned for the study , divided in to three gruops to comparing new combination of prp with prf in management of TMJ OA

ELIGIBILITY:
Inclusion Criteria:

Adult pt with OA

Exclusion Criteria:

Medicaly compromised

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Pain severty | 6 months
  Visual analog scale measure for pain most sever pain take 10 minimum pain take 0

SECONDARY OUTCOMES:
Maximum mouth opening | 6 months
  Measured with calipar

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ab Ghany, Prof, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No